

# Me & You-Tech: A Socio-Ecological Solution to Teen Dating Violence for the Digital Age

NCT05225727

Version Date: 09/16/2022





# Assent Form For Participating in Research Age 7 – 17 Years

**Protocol Title:** Me & You Tech

Principal Investigator: Melissa Peskin, PhD and Ross Shegog, PhD

Study Contact: Andrea Siceluff,

# Invitation to take part in a research study

Drs. Peskin and Shegog are inviting you to take part in a research study. You need to know about the study so you can decide if you would like to join the study or not. If you enter the study you will be asked to sign this form.

Your parents have already agreed that we can talk to you about being in the study. If you want to be in this study, you will be asked to sign this form.

#### Why is this study being done?

We are inviting you to take part in a research study because we are trying to learn more about how to youth, like you, learn skills to have healthy relationships. We want the program to help parents and youth communicate and connect better. The reason we are doing this study is to have kids test part of the digital program and see how well the program helps kids your age have good relationships, and help you speak to your parent about preventing dating violence. This program will also aim to help other adults, such as teachers and counselors, help other kids your age have healthy relationships. The overall outcome we want is to promote healthy relationships and prevent youth dating violence.

#### What will happen if you join the study?

If you agree to be in this study, the following things will happen:

- Participate in three (3) surveys that would take about 25-30 minutes to complete each
  - o Complete a survey before the first lesson to answer some questions about themselves and what they know and think about healthy relationships
  - O Complete a survey at the end of the program to answer some questions again about what they know and think about healthy relationships
  - O Complete a final survey about 9-12 months after the completion of the program about what they know and think about healthy relationships
- Participate in thirteen (13) computer-based modules that last about 25 minutes each
  - Complete questions during the modules
- Complete two (2) questions at the beginning and end of each module about how important and how well they know topics around healthy relationships

You will complete all of the lessons and surveys in school.

## How long will this take?

You total time will be about 8 hours over the course of the program. You will be in this study 8 months.

#### What are the benefits to taking part in this study?

Taking part in this study may or may not help you. Information from this study might help researchers to come up with better prevention programs to help youth have healthy relationships.

Contact Name: Andrea Siceluff
Telephone Number:



# What are some of the risks and discomforts? What could happen that no one would like?

There is very little risk to being in the study. Many middle school children like yourself have used the program on which Me & You Tech is based, but it is possible that you might feel embarrassed by some of the topics. There is always the risk of possible loss of private information. Remember you would not have to take part in any lesson activity that you do not want to.

#### Can you stop being in this study?

Your parent(s) or legal guardian must give permission for you to take part in this study, but you can choose if you want to be in this study or not. You do not have to be in the study. No one will be mad at you if you do not want to do this. If you do not want to be in this study, just tell someone. You do not have to tell them a reason. If you decide to be in the study, you can stop at any time.

# Is there a cost to be in the study?

There is no cost to participate in the study. If you choose to participate in the study, you will be reimbursed \$5.00 gift card when you return your completed consent, \$5.00 gift card for completing the baseline survey, \$5.00 for completing the second survey and \$10.00 gift card for completing the third survey.

## Who will know you are in the study?

When researchers are working on a research project like this, everything you say and everything they write down is private. Researchers don't talk or show the information to anyone who is not working on the study unless you are in danger and need help right away. When anything is written down about you, a special number is written instead of your name. The list and codes of names are kept in a secure locked file.

#### What if you have any questions?

You can ask questions any time. You can ask now or you can ask later. You can talk to the study doctor or you can talk to someone else. If you would like to contact the researcher, she can be contacted at





| Si | gn | at | ur | es |
|----|----|----|----|----|

Sign this paper if you decide you want to volunteer for the study. It is not a promise or contract. It just means that you have read this and that you understand what we are asking. It also means that you would like to try it. Remember that you can always change your mind by just saying so to your parents or anyone working in this study. You understand everything that has been explained to you. You will get a copy of this assent form.

| Printed Name of Subject | | |
|----------------------------------------------|------|------|
| Signature of Subject | Date | Time |
| Printed Name of Individual Obtaining Assent | | |
| Tillited Name of Individual Obtaining Assent | | |
| Signature of Individual Obtaining Assent | Date | Time |

**CPHS STATEMENT:** This study (HSC-SPH-19-0253) has been reviewed by the Committee for the Protection of Human Subjects (CPHS) of the University of Texas Health Science Center at Houston. For any questions about research subject's rights, or to report a research-related injury, call the CPHS at

